CLINICAL TRIAL: NCT00433485
Title: In Vivo and In Vitro Pharmacology of Sirolimus in Subjects With Basal Cell Nevus Syndrome
Brief Title: Topical Sirolimus in Patients With Basal Cell Nevus Syndrome and in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Prevention
Other Study IDs: CDR0000522464; YALE-HIC-26866
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Neoplastic Syndrome; Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; nevoid basal cell carcinoma syndrome
MeSH Terms: conditions — Neoplasms; Carcinoma, Basal Cell; Basal Cell Nevus Syndrome | interventions — Sirolimus; Comparative Genomic Hybridization; Gene Expression Profiling; Microarray Analysis; Mass Spectrometry; Biopsy

INTERVENTIONS:
Drug: sirolimus
Genetic: comparative genomic hybridization
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis
Other: mass spectrometry
Procedure: biopsy

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with basal cell nevus syndrome and from healthy participants in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to basal cell nevus syndrome. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of sirolimus may keep basal cell skin cancer from forming in patients with basal cell nevus syndrome.

PURPOSE: This phase I trial is studying topical sirolimus in patients with basal cell nevus syndrome and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare messenger RNA and protein expression patterns in patients with basal cell nevus syndrome (BCNS) vs in cultured cells of healthy participants (control) before treatment to identify a set of genes that are differentially expressed in BCNS.
* Assess the effects of topical sirolimus on gene expression (genes identified in the primary objective) in vivo using keratinocytes, fibroblasts, and lymphocytes from patients with BCNS and from healthy participants (controls) by targeted expression methods.

OUTLINE: Patients and healthy participants receive topical sirolimus ointment twice daily for 12 weeks.

Blood and skin biopsies are obtained at baseline and at week 12 for gene and protein expression studies. Alterations in RNA are measured by microarray analysis. Alterations in protein expression are measured by 2-dimensional gel electrophoresis and matrix-assisted laser desorption ionization time-of-flight mass spectrometry.

After completion of study therapy, patients and healthy participants are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 16 patients and healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patient

  * Confirmed diagnosis of basal cell nevus syndrome (BCNS)
  * Known patched (PTCH) gene mutation

    * Must have full sequence of coding exons with intron/exon junctions in the PTCH gene OR prior genetic testing confirming PTCH mutation by the Yale University DNA Diagnostics Laboratory
* Age- and sex-matched healthy participant (control)

  * Unaffected relative of patient OR normal healthy volunteer with no family history of BCNS or features of BCNS

    * No unrelated healthy participant meeting any of the following clinical criteria for BCNS:

      * Lamellar calcification of the falx cerebri
      * Prior odontogenic keratocyst or any jaw cyst for which a histopathologic diagnosis cannot be ascertained
      * Palmar or plantar pits typical of BCNS
      * More than 3 basal cell carcinomas (BCC) in a lifetime or 1 BCC under the age of 30
      * History of medulloblastoma
    * No unrelated healthy participant with 2 or more of the following features:

      * History of ovarian or cardiac fibroma
      * Mesenteric or pleural cysts
      * Polydactyly
      * Macrocephaly determined after adjustment for height
      * Craniofacial features of BCNS, including cleft palate, frontal bossing, hypertelorism, iris coloboma or other developmental defects of the eye, or coarse facies
      * Vertebral anomalies, including spina bifida occulta outside the lumbar region
      * Bifid or splayed ribs
      * Other radiographic findings, including bridging of the sella turcica, nonlamellar calcification of the falx cerebri, or flame-shaped lucencies in the phalanges = 1-3 BCCs over the age of 30

PATIENT CHARACTERISTICS:

* WBC ≥ 4,000/mm³
* Neutrophil count ≥ 2,000/mm³
* Platelet count ≥ 150,000/mm³
* Hemoglobin ≥ 11.5 g/dL
* Bilirubin 0.3-1.0 mg/dL
* AST 17-59 U/L
* PTT 10-13 seconds OR INR 1.0-1.4
* Creatinine clearance > 50 mL/min
* Cholesterol < 350 mg/dL
* Triglycerides < 400 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective contraception for ≥ 1 month before, during, and for ≥ 12 weeks after study treatment
* No active infection
* No alcohol or drug abuse
* No psychiatric disorder or mental deficiency that would preclude study compliance
* No uncontrolled hypertension (i.e., blood pressure > 140/90 mm Hg on > 2 measurements)
* No chronic active infection requiring treatment
* No untreated reactive purified protein derivative of tuberculin (PPD)
* No HIV-1 infection
* No infection requiring antibiotics within the past 30 days
* No other skin disease affecting broad areas of the body, including the region to be treated and biopsied
* No known hepatitis B or C infection (detectable RNA off antiviral therapy)
* No immune deficiency disorder
* No known hypersensitivity to sirolimus or macrolide antibiotics (e.g., erythromycin, azithromycin, or clarithromycin)
* No cancer within the past 5 years except basal cell skin cancer

PRIOR CONCURRENT THERAPY:

* At least 1 month since prior investigational drugs
* No concurrent dietary supplements, including Hypericum perforatum (St. John's wort) or megadose vitamins
* No other concurrent immunosuppressive medications, including corticosteroids
* No concurrent medications known to interfere with sirolimus metabolism
* No concurrent anticoagulants
* No concurrent acetylsalicyclic acid or other drugs affecting platelet function or number
* No routine (i.e., > 2 doses/week) use of nonsteroidal anti-inflammatory drugs
* No drugs or substances that would effect sirolimus blood concentrations, including any of the following:

  * Nicardipine
  * Verapamil
  * Clotrimazole
  * Fluconazole
  * Itraconazole
  * Troleandomycin
  * Cisapride
  * Metoclopramide
  * Clarithromycin
  * Erythromycin
  * Bromocriptine
  * Cimetidine
  * Danazol
  * HIV-protease inhibitors (e.g., ritonavir or indinavir)
  * Phenobarbital
  * Carbamazepine
  * Phenytoin
  * Rifabutin
  * Rifapentine
  * Grapefruit juice
  * Vaccinations (especially live vaccines)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Alterations in RNA as measured by microarray analysis
Alterations in protein expression as measured by 2-dimensional gel electrophoresis and matrix-assisted laser desorption ionization time-of-flight mass spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Allen E. Bale, MD, Principal Investigator — Yale University